CLINICAL TRIAL: NCT06051695
Title: A Seamless Phase 1/2 Study to Evaluate the Safety and Efficacy of Mesothelin-Targeting Autologous Logic-gated Tmod™ CAR T Products, in Heterozygous HLA-A*02 Adults With Recurrent Unresectable, Locally Advanced, or Metastatic Solid Tumors That Express MSLN and Have Lost HLA-A*02 Expression
Brief Title: A Study to Evaluate the Safety and Efficacy of Mesothelin-Targeting Logic-gated CAR T, in Participants With Solid Tumors That Express MSLN and Have Lost HLA-A*02 Expression
Acronym: EVEREST-2
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: A2 Biotherapeutics Inc. (Industry)
Collaborators: Tempus AI (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A2B694-101
Record Dates: First submitted 2023-09-18; First posted 2023-09-25 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Solid Tumor, Adult; Colorectal Cancer; NSCLC; Non Small Cell Lung Cancer; NSCLC, Recurrent; Non-Small Cell Squamous Lung Cancer; Pancreas Cancer; Pancreatic Neoplasm; Colorectal Adenocarcinoma; CRC; Colon Cancer; Rectal Cancer; Cancer; Ovarian Cancer; Ovarian Neoplasms; Mesothelioma; Mesothelioma, Malignant; Ovary Cancer; Lung Cancer; MESOM
Keywords: CAR T Cell; Solid Tumors; Autologous; T Cell; Mesothelin; MSLN; HLA-A2; Solid Tumors expressing MSLN; Pancreatic; Cell Therapy; Gene Therapy; blocker; Cancer; PANC; CRC; Colorectal Cancer; Lung Cancer; NSCLC; OVCA; MESOM; Ovarian Cancer; Mesothelioma; Logic-gate
MeSH Terms: conditions — Colorectal Neoplasms; Carcinoma, Non-Small-Cell Lung; Recurrence; Pancreatic Neoplasms; Colonic Neoplasms; Rectal Neoplasms; Neoplasms; Ovarian Neoplasms; Mesothelioma; Mesothelioma, Malignant; Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (2):
- Arm 1: A2B694 (Experimental): Patients receive preconditioning lymphodepletion (PCLD) regimen followed by a single dose of A2B694 intravenously on day 0
  Interventions: Biological: A2B694; Diagnostic Test: xT CDx with HLA-LOH Assay
- Arm 2: A2B543 (Experimental): Patients receive preconditioning lymphodepletion (PCLD) regimen followed by a single dose of A2B543 intravenously on day 0
  Interventions: Biological: A2B543; Diagnostic Test: xT CDx with HLA-LOH Assay

INTERVENTIONS:
Biological: A2B694 — Autologous logic-gated Tmod CAR T cells
  Other Names: Tmod CAR T-cell Therapy
  Arms: Arm 1: A2B694
Biological: A2B543 — Autologous logic-gated Tmod CAR T cells
  Other Names: Tmod CAR T-cell Therapy
  Arms: Arm 2: A2B543
Diagnostic Test: xT CDx with HLA-LOH Assay — An investigational next generation sequencing (NGS) in vitro diagnostic (IVD) medical device

SUMMARY:
The goal of this study is to test autologous logic-gated Tmod™ CAR T-cell products in subjects with solid tumors including colorectal cancer (CRC), pancreatic cancer (PANC), non-small cell lung cancer (NSCLC), ovarian cancer (OVCA), mesothelioma (MESO), and other solid tumors that express mesothelin (MSLN) and have lost HLA-A*02 expression.

The main questions this study aims to answer are:

Phase 1: What is the recommended dose that is safe for patients

Phase 2: Does the recommended dose kill solid tumor cells and protect the patient's healthy cells

Participants will be required to perform study procedures and assessments, and will also receive the following study treatments:

Enrollment and Apheresis in BASECAMP-1 (NCT04981119)

Preconditioning Lymphodepletion (PCLD) Regimen

Tmod CAR T cells at the assigned dose

DETAILED DESCRIPTION:
This is a seamless phase 1/2, multi-center, open-label study that enrolls adults with recurrent unresectable, locally advanced, or metastatic (considered non-curative) CRC, NSCLC, PANC, OVCA, MESO or other solid tumors with MSLN expression. Subjects must be germline HLA-A*02 heterozygous, with tumors that express MSLN and have lost HLA-A*02 expression. This study has two arms: Arm 1 is a study of A2B694 and Arm 2 is a study of A2B543.

The purpose of Phase 1 of this study is to determine the safety and the optimal dose of the Tmod products (after PCLD) in participants with solid tumor disease. The purpose of Phase 2 of this study is to determine the further safety and efficacy (how well it treats the solid tumor disease) of the Tmod products.

The treatment available for these cancers and other solid tumors can be toxic, debilitating, and fatal. In the recurrent unresectable, locally advanced, or metastatic setting, the intent of standard of care treatment is typically palliative rather than curative, and has not changed significantly in several decades. A2 Bio hypothesizes that Tmod CAR T-cell therapy will enable the killing of tumor target cells (those cells that express MSLN and have loss of heterozygosity [LOH] for HLA-A*02 protein). Additionally, normal healthy cells that maintain HLA-A*02 expression and co-express MSLN (eg, lung tissue) will not be targeted due to the blocker portion of the Tmod CAR T cell that acts as a self-regulated safety switch that protects normal tissue from damage. A2 Bio believes this will provide a therapeutic safety window compared to previous solid tumor targeting therapies. This hypothesis will be explored in the study.

Participants for this study must enroll and have their T cells collected (apheresis) in the pre-screening BASECAMP-1 study (NCT04981119). T cells are collected, processed and stored for each participant. Upon disease progression the participant may screen for this study (EVEREST-2) and the participant's T cells are manufactured and then infused following PCLD regimen. There is no time requirement between the studies, and patients may go directly from BASECAMP-1 to EVEREST-2 based on their own disease course.

ELIGIBILITY:
Inclusion Criteria:

Key Inclusion Criteria:

1. Appropriately enrolled in the BASECAMP-1 A2 Biotherapeutics, Inc. study, with tissue demonstrating LOH of HLA-A*02 by NGS (whenever possible from the primary site), successful apheresis and PBMC processing, and with sufficient stored cells available for Tmod CAR T-cell therapy
2. Histologically confirmed recurrent unresectable, locally advanced, or metastatic CRC, NSCLC, PANC, OVCA, MESO, or other solid tumors with MSLN expression. Measurable disease is required with lesions of ≥1.0 cm by CT.
3. Received previous required therapy for the appropriate solid tumor disease as described in the protocol
4. Has adequate organ function as described in the protocol
5. ECOG performance status of 0 to 1
6. Life expectancy of ≥3 months
7. Willing to comply with study schedule of assessments including long term safety follow up

Key Exclusion Criteria:

1. Has disease that is suitable for local therapy or able to receive standard of care therapy that is therapeutic and not palliative
2. Prior allogeneic stem cell transplant
3. Prior solid organ transplant
4. MESO with pleural involvement extending into the peritoneum
5. Cancer therapy within 3 weeks or 3 half lives of infusion
6. Radiotherapy within 28 days of infusion
7. Unstable angina, arrhythmia, myocardial infarction, or any other significant cardiac disease within the last 6 months
8. Any new symptomatic pulmonary embolism (PE) or a deep vein thrombosis (DVT) within 3 months of enrollment. Therapeutic dosing of anticoagulants is allowed for history of PE or DVT if greater than 3 months from time of enrollment, and adequately treated
9. History of interstitial lung disease including drug-induced interstitial lung disease and radiation pneumonitis that requires treatment with prolonged steroids or other immune suppressive agents within 1 year
10. Requires supplemental home oxygen
11. Females of childbearing potential who are pregnant or breastfeeding
12. Subjects, both male and female, of childbearing potential who are not willing to practice birth control from the time of consent through 6 months post infusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 474 (Estimated)
Dates: Start 2024-04-03 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Phase 1: Rate of adverse events and dose limiting toxicities (DLTs) by dose level | From the time of Informed consent until 24 months (2 years) post infusion
  Adverse Events and toxicity will be evaluated according to the Cancer Therapy Evaluation Program Common Terminology Criteria for Adverse Events version (CTCAE) 5.0 (or current version). Cytokine release syndrome (CRS) and immune effector cell-associated neurotoxicity syndrome (ICANS) events will be graded according to the criteria described in the current protocol.
Phase 1: Recommended Phase 2 Dose (RP2D) | 21 days post infusion
  The RP2D will be identified utilizing a BOIN study design in addition to considering safety and biomarker analysis.
Phase 2: The Overall Response Rate (ORR) for patients | 24 months post infusion
  The ORR will be evaluated per RECIST v1.1 and assessed by independent central review.

SECONDARY OUTCOMES:
Persistence of Tmod product | up to 24 months post infusion
  Number of Tmod CAR T cells present as assessed by polymerase chain reaction (PCR) (or similar method) on participant blood samples
Cytokine analysis | up to 24 months post infusion
  Cytokine levels such as interferon-gamma (IFN-γ) and interleukin-6 (IL-6) assessed by cytokine analysis on participant blood samples

CONTACTS AND LOCATIONS:
Overall Officials: John Welch, MD, PhD, Study Director — A2 Biotherapeutics
Locations (12):
- United States (12):
  - Banner Health, Gilbert, Arizona
  - UCSD Moores Cancer Center, La Jolla, California
  - UCLA Medical Center, Los Angeles, California
  - Stanford University, Stanford, California
  - Mayo Clinic, Jacksonville, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Washington University, St Louis, Missouri
  - NYU Langone Medical Center, New York, New York
  - The Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Fred Hutchinson Cancer Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
Study data will be shared within 1 year of study completion.
Supporting Information: CSR
Time Frame: Data will be available within 1 year of the completion of the study, the length of time of availability is to be determined.

REFERENCES:
- [Background] Hamburger AE, DiAndreth B, Cui J, Daris ME, Munguia ML, Deshmukh K, Mock JY, Asuelime GE, Lim ED, Kreke MR, Tokatlian T, Kamb A. Engineered T cells directed at tumors with defined allelic loss. Mol Immunol. 2020 Dec;128:298-310. doi: 10.1016/j.molimm.2020.09.012. Epub 2020 Oct 1. PMID 33012527
- [Background] Hwang MS, Mog BJ, Douglass J, Pearlman AH, Hsiue EH, Paul S, DiNapoli SR, Konig MF, Pardoll DM, Gabelli SB, Bettegowda C, Papadopoulos N, Vogelstein B, Zhou S, Kinzler KW. Targeting loss of heterozygosity for cancer-specific immunotherapy. Proc Natl Acad Sci U S A. 2021 Mar 23;118(12):e2022410118. doi: 10.1073/pnas.2022410118. PMID 33731480
- [Background] Beroukhim R, Mermel CH, Porter D, Wei G, Raychaudhuri S, Donovan J, Barretina J, Boehm JS, Dobson J, Urashima M, Mc Henry KT, Pinchback RM, Ligon AH, Cho YJ, Haery L, Greulich H, Reich M, Winckler W, Lawrence MS, Weir BA, Tanaka KE, Chiang DY, Bass AJ, Loo A, Hoffman C, Prensner J, Liefeld T, Gao Q, Yecies D, Signoretti S, Maher E, Kaye FJ, Sasaki H, Tepper JE, Fletcher JA, Tabernero J, Baselga J, Tsao MS, Demichelis F, Rubin MA, Janne PA, Daly MJ, Nucera C, Levine RL, Ebert BL, Gabriel S, Rustgi AK, Antonescu CR, Ladanyi M, Letai A, Garraway LA, Loda M, Beer DG, True LD, Okamoto A, Pomeroy SL, Singer S, Golub TR, Lander ES, Getz G, Sellers WR, Meyerson M. The landscape of somatic copy-number alteration across human cancers. Nature. 2010 Feb 18;463(7283):899-905. doi: 10.1038/nature08822. PMID 20164920
- [Background] Tokatlian T, Asuelime GE, Mock JY, DiAndreth B, Sharma S, Toledo Warshaviak D, Daris ME, Bolanos K, Luna BL, Naradikian MS, Deshmukh K, Hamburger AE, Kamb A. Mesothelin-specific CAR-T cell therapy that incorporates an HLA-gated safety mechanism selectively kills tumor cells. J Immunother Cancer. 2022 Jan;10(1):e003826. doi: 10.1136/jitc-2021-003826. PMID 35091455
- See also: A2 Biotherapeutics Inc. — http://www.a2bio.com